CLINICAL TRIAL: NCT04948229
Title: Annexin A1 as a Potential Prognostic Biomarker for COVID-19 Disease: Case-Control Study
Brief Title: Annexin A1 Levels in SARS-CoV-2 Infection
Status: Completed | Type: Observational
Sponsor: Kafkas University (Other)
Collaborators: Aylin Koseler (Unknown)
Responsible Party: Principal Investigator, Ramazan Sbirli, Dr., Kafkas University
Other Study IDs: Clinical-5
Record Dates: First submitted 2021-06-29; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Annexin A1; Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum analysis will be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: This group will be included subjects who had no history or diagnosis of any disease, no infection history within last two weeks, no history of any particular medication, who were admitted to emergency department (ED) with complaints other than infectious issues, and who gave their written consent to participate in the study.
  Interventions: Other: Blood serum samples
- Moderate Disease Group: This group will be consisted of the patients whose diagnoses of moderate COVID-19 infection were confirmed by positive RT-PCR in ED according to WHO guidelines and who gave their written consent were included in the study.
  Interventions: Other: Blood serum samples
- Severe/Critical Disease Group: This group will be consisted of the patients whose diagnoses of severe/critical COVID-19 infection were confirmed by positive RT-PCR in ED according to WHO guidelines and who gave their written consent were included in the study.
  Interventions: Other: Blood serum samples

INTERVENTIONS:
Other: Blood serum samples — Blood serum samples will be taken.

SUMMARY:
The present study aims to determine the clinical predictivity value of blood AnxA1 levels in patients with mild and severe/critical pneumonia induced by COVID-19 and to reveal the alterations of blood AnxA1 levels in patients with pneumonia compared to the control group.The present study is a prospective case-control study, and the required ethics approval was obtained from the Ethics Committee of Pamukkale University (Numbered: E-60116787-020-15062). The study was conducted at Ankara Training and Research Hospital between 10.02.2021 and 15.03.2021. All procedures will carried out on patients were in compliance with the Helsinki Declaration.Study groups were established according to the inclusion and exclusion criteria. Patients whose diagnoses were clinically confirmed as COVID-19 infection according to World Health Organization (WHO) guidelines using a positive reverse transcriptase polymerase chain reaction (RT-PCR) test will be included in the study (15). Individuals will be grouped in the moderate COVID-19 disease group (N=42), severe/critical COVID-19 disease group (N=32), and the healthy control group (N=50).

Healthy group will be included subjects who had no history or diagnosis of any disease, no infection history within last two weeks, no history of any particular medication, who were admitted to emergency department (ED) with complaints other than infectious issues, and who gave their written consent to participate in the study.

Venous blood samples that will be taken when the patients were admitted to ED were withdrawn into a dry test tube that did not contain anti-coagulant and were then centrifugated for 10 minutes at 4000 rpm. Serum samples will be obtained from centrifugation were collected for laboratory analysis. Serum AnxA1 levels were analyzed using a commercially available AnxA1 ELISA Kit (Elabscience, E-EL-H5512, USA), per the manufacturer's protocol.

DETAILED DESCRIPTION:
The present study aims to determine the clinical predictivity value of blood AnxA1 levels in patients with mild and severe/critical pneumonia induced by COVID-19 and to reveal the alterations of blood AnxA1 levels in patients with pneumonia compared to the control group.The present study is a prospective case-control study, and the required ethics approval was obtained from the Ethics Committee of Pamukkale University (Numbered: E-60116787-020-15062). The study was conducted at Ankara Training and Research Hospital between 10.02.2021 and 15.03.2021. All procedures will carried out on patients were in compliance with the Helsinki Declaration.Study groups were established according to the inclusion and exclusion criteria. Patients whose diagnoses were clinically confirmed as COVID-19 infection according to World Health Organization (WHO) guidelines using a positive reverse transcriptase polymerase chain reaction (RT-PCR) test will be included in the study (15). Individuals will be grouped in the moderate COVID-19 disease group (N=42), severe/critical COVID-19 disease group (N=32), and the healthy control group (N=50).

Healthy group will be included subjects who had no history or diagnosis of any disease, no infection history within last two weeks, no history of any particular medication, who were admitted to emergency department (ED) with complaints other than infectious issues, and who gave their written consent to participate in the study.

Venous blood samples that will be taken when the patients were admitted to ED were withdrawn into a dry test tube that did not contain anti-coagulant and were then centrifugated for 10 minutes at 4000 rpm. Serum samples will be obtained from centrifugation were collected for laboratory analysis. Serum AnxA1 levels were analyzed using a commercially available AnxA1 ELISA Kit (Elabscience, E-EL-H5512, USA), per the manufacturer's protocol.

Inclusion Criteria Patient Groups: Patients whose diagnoses of COVID-19 infection were confirmed by positive RT-PCR in ED according to WHO guidelines and who gave their written consent were included in the study (15).

Control Group: Subjects with no history of a known disease, no infectious symptoms, no drug use, and who provided written consent were included in the study.

ELIGIBILITY:
Healthy Group

Inclusion Criteria:

* Not to have any known disease
* Not to use any drugs
* Not to have any history of chronic disease and infection
* Not to have any infectious symptoms
* To give informed consent.

Exclusion Criteria:

* To have any known disease
* To use any drugs Moderate Disease Group

Inclusion Criteria:

* To have confirmed COVID-19 infection
* To have positive RT-PCR in ED according to WHO guidelines
* To give informed consent.

Exclusion Criteria:

* To have any heart, kidney or liver failure
* To have acute pulmonary embolism
* To have deep venous thrombosis or chronic inflammatory disease
* To have pregnancy

Severe/Critical Disease Group

Inclusion Criteria:

* To have confirmed severe/critical COVID-19 infection
* To have positive RT-PCR in ED according to WHO guidelines
* To give informed consent.

Exclusion Criteria:

* To have any heart, kidney or liver failure
* To have acute pulmonary embolism
* To have deep venous thrombosis or chronic inflammatory disease
* To have pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects will be included in the present study were clinically evaluated using WHO diagnosis and treatment guidelines for COVID-19. The patient management algorithms will be administered due to the updates of these guidelines. The patient groups will be categorized as moderate disease and severe/critical disease according to WHO guidelines. Individuals will be grouped in the moderate COVID-19 disease group (N=42), severe/critical COVID-19 disease group (N=32), and the healthy control group (N=50).
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
To determine differences between controls and patients groups in terms of serum Annexin A1 levels | 15 days
  Serum annexin A1 levels will be analysed statistically and the differences will be determined between the patients and controls.

SECONDARY OUTCOMES:
To determine differences between moderate and severe/critical disease groups in terms of serum Annexin A1 levels. | 17 days
  Serum annexin A1 levels will be analysed statistically and the differences will be determined between the moderate and severe/critical disease group

CONTACTS AND LOCATIONS:
Locations (1):
- Ramazan Sabirli, Kars, Outside of the US, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No